CLINICAL TRIAL: NCT07243327
Title: A Prospective Randomized Controlled Trial Comparing the Effectiveness of Extracorporeal Shockwave Therapy and Conventional Physical Therapy in Patients With Greater Trochanteric Pain Syndrome
Brief Title: ESWT vs Conventional Physical Therapy in Greater Trochanteric Pain Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Zeynep Karakuzu Güngör, Kanuni Sultan Suleyman Training and Research Hospital, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTAS-ESWT-2025-01
Record Dates: First submitted 2025-11-14; First posted 2025-11-21 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Greater Trochanteric Pain Syndrome
Keywords: Extracorporeal shockwave therapy; Physical therapy; Hip pain; ESWT
MeSH Terms: interventions — Extracorporeal Shockwave Therapy; Transcutaneous Electric Nerve Stimulation; High-Energy Shock Waves

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel-group, randomized controlled trial (1:1 allocation).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESWT Group (Experimental): Extracorporeal shockwave therapy applied 5 sessions over 3 weeks (15 Hz, 3 bar, 2000 pulses). Standard hip exercises included.
  Interventions: Device: Extracorporeal Shockwave Therapy (ESWT)
- Conventional Physical Therapy Group (Active Comparator): 10 sessions of TENS (20 min), hot pack (20 min), and continuous ultrasound (1.5 W/cm², 5 min). Standard hip exercises included.
  Interventions: Other: TENS; Hot Pack; Ultrasound

INTERVENTIONS:
Device: Extracorporeal Shockwave Therapy (ESWT) — ESWT applied with Elmed Vibrolith Ortho device at 15 Hz, 3 bar, 2000 pulses, 5 sessions over 3 weeks.
  Arms: ESWT Group
Other: TENS; Hot Pack; Ultrasound — 10 sessions of TENS (20 min), hot pack (20 min), and continuous ultrasound (1.5 W/cm², 5 min).
  Arms: Conventional Physical Therapy Group

SUMMARY:
This study aims to compare the effectiveness of Extracorporeal Shockwave Therapy (ESWT) with conventional physical therapy in patients with Greater Trochanteric Pain Syndrome (GTPS). GTPS is a common cause of lateral hip pain, often related to gluteal tendinopathy rather than trochanteric bursitis. Sixty patients will be randomly assigned to two groups: ESWT or conventional physical therapy (TENS, hot pack, ultrasound). Pain (VAS), hip function (Harris Hip Score), lower limb function (LEFS), and global improvement will be evaluated at baseline, week 3, and week 12. The purpose of this study is to determine which treatment provides greater pain relief and functional improvement.

DETAILED DESCRIPTION:
Greater Trochanteric Pain Syndrome (GTPS) is a frequent cause of lateral hip pain and is now understood to be primarily associated with gluteus medius and minimus tendinopathy rather than inflammation of the trochanteric bursa. Although several conservative treatments are available, including nonsteroidal anti-inflammatory drugs and physical therapy modalities, there is no consensus on the most effective treatment strategy. Extracorporeal Shockwave Therapy (ESWT) has emerged as a potential non-invasive treatment option that may promote tissue regeneration, reduce pain, and improve tendon healing.

This prospective randomized controlled trial will include 60 patients aged 18-65 years with MRI-confirmed GTPS. Participants will be randomly assigned (1:1) to either the ESWT group or the conventional physical therapy group. The ESWT group will receive five sessions over 3 weeks (15 Hz, 3 bar, 2000 pulses). The physical therapy group will receive 10 sessions of TENS (20 minutes), hot pack (20 minutes), and continuous ultrasound (1.5 W/cm², 5 minutes). Both groups will be given a standardized exercise program.

Outcome measures include the Visual Analog Scale (VAS) for pain (night, rest, activity), Harris Hip Score, Lower Extremity Functional Scale (LEFS), and the Global Rating of Change Scale. Assessments will be performed at baseline, week 3, and week 12. The primary objective is to compare the effect of ESWT versus conventional physical therapy on pain reduction. Secondary objectives include evaluating functional improvements and global patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Lateral hip pain for at least 3 months
* Ability to understand study procedures and provide informed consent

Exclusion Criteria:

* Hip deformities
* Gluteus medius, gluteus minimus, or piriformis tendon tears
* Lumbar radiculopathy or history of lumbar spine surgery
* Recent trauma or active infection in the hip region
* Corticosteroid injection to the hip within the last 6 months
* Neurological, psychiatric, or rheumatologic diseases
* Active malignancy or systemic inflammatory disease
* Cognitive impairment preventing cooperation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analog Scale (VAS) Pain Score | Baseline, Week 3, and Week 12
  Pain intensity will be assessed using a 0-10 Visual Analog Scale (VAS) for activity, rest, and night pain. The primary endpoint is the change in VAS score from baseline to Week 12.

SECONDARY OUTCOMES:
Harris Hip Score | Baseline, Week 3, and Week 12
  Hip function will be evaluated using the Harris Hip Score, which includes pain, daily activities, gait, and range of motion parameters. Higher scores indicate better hip function.
Lower Extremity Functional Scale (LEFS) | Baseline, Week 3, and Week 12
  The LEFS questionnaire will be used to assess lower limb function. It consists of 20 items scored from 0 to 4 (total score 0-80), with higher scores indicating better function.
Global Rating of Change (GROC) | Week 3 and Week 12
  Overall patient-perceived improvement will be assessed using the Global Rating of Change Scale, scored from -1 (worse) to +3 (near normal improvement).

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Karakuzu Güngör, Principal Investigator — Kanuni Sultan Suleyman Training and Research Hospital
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No